CLINICAL TRIAL: NCT01067963
Title: Self-management of Type 2 Diabetes and Chronic Kidney Disease
Brief Title: Self-Management and Resourceful Transition of Type 2 Diabetes With Stage 3 Kidney Disease
Acronym: SMaRT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Robert Wood Johnson Foundation (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-0939; 1UL1RR025780 (NIH); RWJ64198 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic
Keywords: self-care; self-management; health behavior change; motivational interviewing; computer assisted learning
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral-education/counseling (Experimental): Computer assisted education and telephone counseling using motivational interviewing.
  Computer assisted education and motivational interviewing
  Interventions: Behavioral: Computer assisted education and motivational interviewing.
- Group talks/social chat (Placebo Comparator): Group session talks on general topics about healthy lifestyle, printed power point handouts, telephone calls comprised of social conversation to discuss the handout content.
  Interventions: Behavioral: Group talks/social chat

INTERVENTIONS:
Behavioral: Computer assisted education and motivational interviewing. — 9 study contact points. 3-week intervention using computer-assisted learning modules and telephone counseling using motivational interviewing.
  Other Names: Experimental Group
  Arms: Behavioral-education/counseling
Behavioral: Group talks/social chat — 9 study contact points. 3 group talk session on general topics about healthy lifestyle, printed power point handouts, telephone calls comprised of social conversation to discuss the handout content.
  Other Names: Attention Control Group
  Arms: Group talks/social chat

SUMMARY:
The purpose of this study is to establish the usefulness and the impact of a tailored behavioral-education and counseling intervention titled Self-Management and Resourceful Transition (S.M.a.R.T) among patients with type 2 diabetes mellitus and stage 3 chronic kidney disease, in order to help them to manage their behaviors related to their condition and health.

DETAILED DESCRIPTION:
The SMaRT intervention is a 3-week intervention that uses a combined behavioral-education and counseling methodology. The combined intervention involves computer-aided education alongside telephone counseling via motivational interviewing. The computer-aided education is tailored to the diagnoses of type 2 diabetes and chronic kidney disease and designed in a learning module approach to facilitate goal-setting and discussion of health concerns with greater efficacy and in a more informed way during the brief office visit. Such Computer-aided education has been used to improve diabetes self-management and glycemic control in middle-aged to older adults with moderate success. The inclusion of CKD information will augment current diabetes self-management intervention. The telephone counseling using the evidence-based behavioral change approach of motivational interviewing is a patient-centered approach of partnering with patients by eliciting their health-related concerns. This approach tailors the SMaRT intervention to include collaborative goal-setting with guidance based upon the patient's readiness for change.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Type 2 Diabetes
* 18-85 years old
* Stage 3 Chronic Kidney Disease
* Speaks and reads English

Exclusion Criteria:

* Hypoglycemia with 3rd party treatment in past 3 months
* Type 1 Diabetes
* On Dialysis
* Does not speak English
* Factors likely to preclude protocol adherence

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Primary outcomes utilized in this study will be disease burden (measured as diabetes-related distress), quality of life (measured as health related QOL), and glycemic health (measured as hemoglobin A1C). | One year

SECONDARY OUTCOMES:
Secondary exploratory outcomes for quality of life include measures of health-related quality of life for diabetes and overall quality of life. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J. Sakraida, PhD, RN, Principal Investigator — University of Colorado Denver College of Nursing; Alkesh Jani, MD, Principal Investigator — University of Colorado Denver, School of Medicine and VA Eastern Colorado Hospital
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - VA Eastern Colorado Hospital, Denver, Colorado

REFERENCES:
- [Background] Coresh J, Astor BC, Greene T, Eknoyan G, Levey AS. Prevalence of chronic kidney disease and decreased kidney function in the adult US population: Third National Health and Nutrition Examination Survey. Am J Kidney Dis. 2003 Jan;41(1):1-12. doi: 10.1053/ajkd.2003.50007. PMID 12500213
- [Background] Franz MJ, Bantle JP, Beebe CA, Brunzell JD, Chiasson JL, Garg A, Holzmeister LA, Hoogwerf B, Mayer-Davis E, Mooradian AD, Purnell JQ, Wheeler M; American Diabetes Association. Evidence-based nutrition principles and recommendations for the treatment and prevention of diabetes and related complications. Diabetes Care. 2003 Jan;26 Suppl 1:S51-61. doi: 10.2337/diacare.26.2007.s51. No abstract available. PMID 12502619
- [Background] Berridge E, Roudsari A, Taylor S, Carey S. Computer-aided learning for the education of patients and family practice professionals in the personal care of diabetes. Comput Methods Programs Biomed. 2000 Jul;62(3):191-204. doi: 10.1016/s0169-2607(00)00067-5. PMID 10837906
- [Background] National Kidney Foundation [NKF]. Kidney disease outcomes quality initiative (K/DOQI): Clinical Practice Guideline 2-evaluation and treatment 2002: Accessed March 21, 2008 from http://www.kidney.org/professionals/kdoqi/guidelines_ckd/p4_class_g2.htm.
- [Background] Khosla N, Bakris G. Lessons learned from recent hypertension trials about kidney disease. Clin J Am Soc Nephrol. 2006 Mar;1(2):229-35. doi: 10.2215/CJN.00840805. Epub 2005 Nov 30. No abstract available. PMID 17699211
- [Background] Kshirsagar AV, Joy MS, Hogan SL, Falk RJ, Colindres RE. Effect of ACE inhibitors in diabetic and nondiabetic chronic renal disease: a systematic overview of randomized placebo-controlled trials. Am J Kidney Dis. 2000 Apr;35(4):695-707. doi: 10.1016/s0272-6386(00)70018-7. PMID 10739792
- [Background] National Kidney Foundation [NKF]. Kidney Disease Outcomes Quality Initiative (K/DOQI): Clinical Practice Guideline 9-assoc of level of GFR with nutritional status and Guideline 24-dietary protein intake for nondialyzed patients, 2002.
- [Background] Perlman RL, Kiser M, Finkelstein F, Eisele G, Roys E, Liu L, Burrows-Hudson S, Port F, Messana JM, Bailie G, Rajagopalan S, Saran R. The longitudinal chronic kidney disease study: a prospective cohort study of predialysis renal failure. Semin Dial. 2003 Nov-Dec;16(6):418-23. doi: 10.1046/j.1525-139x.2003.16093.x. PMID 14629599
- [Background] KDOQI. KDOQI Clinical Practice Guidelines and Clinical Practice Recommendations for Diabetes and Chronic Kidney Disease. Am J Kidney Dis. 2007 Feb;49(2 Suppl 2):S12-154. doi: 10.1053/j.ajkd.2006.12.005. No abstract available. PMID 17276798
- [Background] Glasgow RE, Hiss RG, Anderson RM, Friedman NM, Hayward RA, Marrero DG, Taylor CB, Vinicor F. Report of the health care delivery work group: behavioral research related to the establishment of a chronic disease model for diabetes care. Diabetes Care. 2001 Jan;24(1):124-30. doi: 10.2337/diacare.24.1.124. PMID 11194217
- [Background] Rollnick S, Mason P, Butler C. Health behavior change: A guide for practitioners. Edinburgh, Scotland: Churchill Livingstone Elsevier; 1999.
- [Background] Prochaska JO, DiClemente CC. Stages of change in the modification of problem behaviors. Prog Behav Modif. 1992;28:183-218. No abstract available. PMID 1620663
- [Background] Rollnick S, Miller WR, Butler CC. Motivational interviewing in health care: Helping patients change behavior. New York: Guilford Press; 2007.
- [Background] Glasgow RE, Boles SM, McKay HG, Feil EG, Barrera M Jr. The D-Net diabetes self-management program: long-term implementation, outcomes, and generalization results. Prev Med. 2003 Apr;36(4):410-9. doi: 10.1016/s0091-7435(02)00056-7. PMID 12649049
- [Background] Gerber BS, Brodsky IG, Lawless KA, Smolin LI, Arozullah AM, Smith EV, Berbaum ML, Heckerling PS, Eiser AR. Implementation and evaluation of a low-literacy diabetes education computer multimedia application. Diabetes Care. 2005 Jul;28(7):1574-80. doi: 10.2337/diacare.28.7.1574. PMID 15983303
- [Background] Hettema J, Steele J, Miller WR. Motivational interviewing. Annu Rev Clin Psychol. 2005;1:91-111. doi: 10.1146/annurev.clinpsy.1.102803.143833. PMID 17716083
- [Background] Brown SA. Studies of educational interventions and outcomes in diabetic adults: a meta-analysis revisited. Patient Educ Couns. 1990 Dec;16(3):189-215. doi: 10.1016/0738-3991(90)90070-2. PMID 2149753
- [Background] Himmelfarb J. Chronic kidney disease and the public health: gaps in evidence from interventional trials. JAMA. 2007 Jun 20;297(23):2630-3. doi: 10.1001/jama.297.23.2630. No abstract available. PMID 17579231
- [Background] American Diabetes Association. Standards of medical care in diabetes--2008. Diabetes Care. 2008 Jan;31 Suppl 1:S12-54. doi: 10.2337/dc08-S012. No abstract available. PMID 18165335
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Sakraida TJ, Robinson MV. Health literacy self-management by patients with type 2 diabetes and stage 3 chronic kidney disease. West J Nurs Res. 2009 Aug;31(5):627-47. doi: 10.1177/0193945909334096. Epub 2009 Apr 23. PMID 19390053
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Hays RD, Kallich JD, Mapes DL, Coons SJ, Carter WB. Development of the kidney disease quality of life (KDQOL) instrument. Qual Life Res. 1994 Oct;3(5):329-38. doi: 10.1007/BF00451725. PMID 7841967
- [Background] Bradley C, Todd C, Gorton T, Symonds E, Martin A, Plowright R. The development of an individualized questionnaire measure of perceived impact of diabetes on quality of life: the ADDQoL. Qual Life Res. 1999;8(1-2):79-91. doi: 10.1023/a:1026485130100. PMID 10457741
- [Background] Ware J, Snow K, Kosinski M, Gandek B. SF-36 Health Survey: Manual and Interpretation Guide. Boston: The Health Institute, New England Medical Centre;1993.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Woodcock AJ, Julious SA, Kinmonth AL, Campbell MJ; Diabetes Care From Diagnosis Group. Problems with the performance of the SF-36 among people with type 2 diabetes in general practice. Qual Life Res. 2001;10(8):661-70. doi: 10.1023/a:1013837709224. PMID 11871587
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Kavookjian J, Berger B, Anderson-Harper H, Barker K, Grimley D, Pearson R, et al. The relationship between readiness for diabetes self-care and glycemic control: The development of a diagnostic tool for pharmacist intervention. Journal of American Pharmaceutical Association 41:320, 2001.
- [Background] Greene GW, Rossi SR, Rossi JS, Velicer WF, Fava JL, Prochaska JO. Dietary applications of the stages of change model. J Am Diet Assoc. 1999 Jun;99(6):673-8. doi: 10.1016/S0002-8223(99)00164-9. No abstract available. PMID 10361528
- [Background] Hellsten LA, Nigg C, Norman G, Burbank P, Braun L, Breger R, Coday M, Elliot D, Garber C, Greaney M, Lees F, Matthews C, Moe E, Resnick B, Riebe D, Rossi J, Toobert D, Wang T. Accumulation of behavioral validation evidence for physical activity stage of change. Health Psychol. 2008 Jan;27(1S):S43-53. doi: 10.1037/0278-6133.27.1(Suppl.).S43. PMID 18248105
- [Background] Greene GW, Rossi SR, Reed GR, Willey C, Prochaska JO. Stages of change for reducing dietary fat to 30% of energy or less. J Am Diet Assoc. 1994 Oct;94(10):1105-10; quiz 1111-2. doi: 10.1016/0002-8223(94)91127-4. PMID 7930314
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Stanford Patient Education Research Center, Self Efficacy for Diabetes. Stanford (Accessed March 28, 2008, at http://patienteducation.stanford.edu/research/sediabetes.html.)
- [Background] National Kidney Foundation [NKF]. Kidney disease outcomes quality initiative (K/DOQI): Clinical practice Guideline 4-Estimation of GFR Part 5 evaluation of laboratory measures for clinical assessment of kidney disease. 2002: Accessed March 27, 2008 from http://www.kidney.org/professionals/kdoqi/guidelines_ckd/p5_lab_g4.htm.
- [Background] Lynn MR. Determination and quantification of content validity. Nurs Res. 1986 Nov-Dec;35(6):382-5. No abstract available. PMID 3640358
- [Background] Sheiner LB, Rubin DB. Intention-to-treat analysis and the goals of clinical trials. Clin Pharmacol Ther. 1995 Jan;57(1):6-15. doi: 10.1016/0009-9236(95)90260-0. No abstract available. PMID 7828382
- [Background] Aubert RE, Herman WH, Waters J, Moore W, Sutton D, Peterson BL, Bailey CM, Koplan JP. Nurse case management to improve glycemic control in diabetic patients in a health maintenance organization. A randomized, controlled trial. Ann Intern Med. 1998 Oct 15;129(8):605-12. doi: 10.7326/0003-4819-129-8-199810150-00004. PMID 9786807